CLINICAL TRIAL: NCT04813913
Title: VASCular Impact of Angiogenic Treatment in Patients With Advanced Colorectal Cancer
Acronym: VASCATAQ
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/0184 HP
Record Dates: First submitted 2020-06-25; First posted 2021-03-24 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Oncology
MeSH Terms: conditions — Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- bevacizumab (Experimental): bevacizumab in combination with IV fluoropyrimidine chemotherapy.
  Interventions: Drug: Bevacizumab in combination with chemotherapy based on fluoropyrimidine IV

INTERVENTIONS:
Drug: Bevacizumab in combination with chemotherapy based on fluoropyrimidine IV — Enrollement of major patient with colorectal cancer of the adenocarcinoma type, stage IV, histologically confirmed, naive in antineoplastic treatment and eligible to start a systemic carcinological treatment comprising bevacizumab in combination with chemotherapy based on fluoropyrimidine IV. The main objective is to show that there is an increase in the stiffness of the carotid artery at 4 months in patients with stage IV colorectal cancer exposed to bevacizumab.

SUMMARY:
Antiangiogenic treatments are used in many tumor locations such as metastatic colorectal cancer (mCRC) with a significant improvement in carcinological results on overall survival and / or progression-free survival. However, their use is characterized by an increase in side effects and in particular cardiovascular effects such as high blood pressure (hypertension). One of the main classes of antiangiogens used in this indication is that of monoclonal antibodies, the leader of which is bevacizumab (Avastin®, Roche, Bale, Switzerland). Bevacizumab works by inhibiting endothelial vascular growth factor-dependent neoangiogenesis (vascular endothelial growth factor VEGF). In the reference studies, the inhibition of VEGF, whether extracellular (monoclonal antibody directed against VEGFA) or intracellular (receptor inhibitors with tyrosine kinase activity), induces hypertension of all grades, observed in 25% to 40 % of patients including 8 to 17% of severe grades (≥ grade 3 NCI-CTCAE). In terms of pathophysiology, inhibition of VEGFA results in a decrease in the availability of nitric oxide (NO) at the endothelial level and the appearance of arteriolar rarefaction. This induces an increase in peripheral resistance responsible ultimately for an increase in blood pressure. The occurrence of hypertension induced by anti-VEGF treatment seems to be predictive of the carcinological response in certain oncological situations such as metastatic breast cancer9, glioblastoma and mRCC. Furthermore, it has also been shown that there is an early attack on the elastic conductance arteries (branches of the aorta and its main ones) characterized by an increase in their rigidity in patients exposed to a VEGF receptor inhibitor with tyrosine activity. kinase or bevacizumab. This increase, whose poor prognostic impact is known at the cardiovascular level is largely independent of the rise in blood pressure and reflects a direct toxicity of treatments at the level of the artery wall. This increase in rigidity, refused when the pressure rises, would be predictive of a low carcinological response rate at 6 months. However, these data are based on populations that are heterogeneous in terms of carcinology and the position prior to or concomitant with other antineoplastic treatments.

In this context, the evaluation of arterial stiffness in the same patient population would make it possible to better define the involvement of the conductive arteries in a clearly defined clinical situation. Joint measurements of the plasma concentration of the treatment as well as those of factors derived from the endothelium and circulating tumor markers which, to our knowledge, have never been carried out in these patients, would make it possible to better specify the mechanisms of involvement and the links between exposure, arterial toxicity and carcinologic efficacy of bevacizumab. Of course, in order to assess more precisely the inherent impact of chemotherapy on the conductance arteries, the evolution of arterial stiffness must take into account the possible effects in patients receiving, for essentially clinical and biological reasons, systemic treatment without antiangiogenic.

ELIGIBILITY:
Inclusion Criteria:

* Patient at least 18 years old,
* Patient with colorectal cancer of the adenocarcinoma type, stage IV, histologically confirmed, mutated or wild tumor RAS status (exons 2, 3 and 4 of the KRAS and NRAS genes), mutated or wild BRAF status, naive in antineoplastic treatment
* Patient eligible to start systemic carcinological treatment including bevacizumab in combination with chemotherapy based on IV fluoropyrimidine,
* General condition WHO grade less than or equal to 3,
* Life expectancy greater than 4 months,
* Patient who has read and understood the information letter and signed the consent form,
* Patient affiliated to a social security scheme,
* Effective contraception (see WHO definition) in women of childbearing age (negative pregnancy test). For postmenopausal women, a confirmatory diagnosis should be obtained (amenorrhea not medically induced for at least 12 months before the inclusion visit).

Exclusion Criteria:

* Previous exposure to anti-VEGF,
* Exposure to treatment for metastatic disease in the 12 months prior to inclusion,
* Other histologically proven neoplasia not considered in complete remission or considered in complete remission for less than two years,
* Bilateral carotid breath,
* Absence of peripheral pulse of the two upper limbs,
* Contraindication to AVASTIN 25 mg / ml concentrate for solution for infusion:

  * Hypersensitivity to the active substance or to any of the excipients,
  * Hypersensitivity to Chinese hamster ovarian cell products or other human or humanized recombinant antibodies,
* Patients:

  * having undergone a major surgical intervention in the 28 days preceding the inclusion or as long as the surgical wound is not completely healed,
  * Unhealed ulcer or wound,
  * having uncontrolled pre-existing hypertension (PAS> or = 170 mm Hg after three repeated measurements at rest),
  * having a history of arterial thromboembolism (transient ischemic attack (TIA), cardiovascular accident (stroke) or recent (<6 months) and / or symptomatic myocardial infarction (MI)
  * having had an invasive dental procedure in the 28 days preceding inclusion,
  * with known proteinuria> 2g / 24h or in whom proteinuria> 2g / 24h is discovered in the case of a positive urine strip 3+ for proteins (excluding urinary tract infection),
  * on aspirin> 325 mg / d,
  * with a colonic prosthesis in place,
* Systemic treatment with anti-EGFR monoclonal antibodies,
* Presence or history of lymphedema of the bilateral upper limbs,
* Patient with poor understanding of spoken or written French,
* Patient deprived of liberty by an administrative or judicial decision or patient placed under the protection of justice, under guardianship or curatorship,
* Pregnant or lactating woman or wishing to breastfeed within 6 months after the last administration of the treatment,
* Patient participating in another drug trial / having participated in another drug trial within 30 days of inclusion,
* History of illness or psychological or sensory abnormality likely to prevent the subject from fully understanding the conditions required for his participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-05-05 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-07-21 (Actual)

PRIMARY OUTCOMES:
Difference in carotid stiffness between baseline and at 4 months of bevacizumab treatment. | Through study completion, an average of 4 months
  Difference in carotid stiffness estimated by the delta of the pulse wave velocity calculated by an applanation tonometry and an ultrasound at the level of the common carotid artery, between baseline and at 4 months of bevacizumab treatment.

SECONDARY OUTCOMES:
Difference of central arterial pressures between baseline and at 4 months of bevacizumab treatment | Through study completion, an average of 4 months
  Differences of central arterial pressures, of aortic stiffness, calculated by a flattening tonometry between the values before exposure and at 4 months of exposure to bevacizumab. Differences between the distensibility of the common carotid artery, calculated from the carotid diameters during the heart beat and estimated by carotid echotracking before, at 4 months of bevacizumab treatment
Difference of central arterial pressures between baseline and at 1 month of bevacizumab treatment | 1 month
  Differences of central arterial pressures, of aortic stiffness, calculated by a flattening tonometry between the values before exposure and at 1 month of exposure to bevacizumab. Differences between the distensibility of the common carotid artery, calculated from the carotid diameters during the heart beat and estimated by carotid echotracking before, at 1 month of bevacizumab treatment
Difference of peripheral arterial pressures between baseline and at 4 months of bevacizumab treatment | 4 months
  Differences of peripheral arterial pressures, of aortic stiffness, calculated by a flattening tonometry between the values before exposure and at 4 months of exposure to bevacizumab. Differences between the distensibility of the common carotid artery, calculated from the carotid diameters during the heart beat and estimated by carotid echotracking before, at 4 months of bevacizumab treatment
Difference of peripheral arterial pressures between baseline and at 1 month of bevacizumab treatment | 1 month
  Differences of peripheral arterial pressures, of aortic stiffness, calculated by a flattening tonometry between the values before exposure and at 1 month of exposure to bevacizumab. Differences between the distensibility of the common carotid artery, calculated from the carotid diameters during the heart beat and estimated by carotid echotracking before, at 1 month of bevacizumab treatment
The evolution of circulating concentrations of markers of endothelial function (nitric oxide [NO], epoxyeicosatrienoic acids [EETs], sVE-cadherin), | 1 and 4 months
  Differences in plasma concentrations of NO, EETs and sVE-cadherin before exposure and at 1 and 4 months of bevacizumab treatment.
Changes in the concentrations of bevacizumab and its autoantibody, of a circulating tumor marker, circulating markers of hypoxia and angiogenesis (HIF1alpha, sVEGFR2, VEGF-A) and their correlations with the proportion of responders, | 12 months
  Correlations between all of these parameters and the proportion of responder or stable patients at 12 months. A patient is considered to be responder or stable or without progression if there is neither a CT argument according to RECIST 1.1 criteria, nor a clinical argument for tumor progression.
Progression-free survival at 12 months. | 12 months
  12-month progression-free survival.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de ROUEN, Rouen, France